CLINICAL TRIAL: NCT00163137
Title: Double-Blind Placebo-Controlled Trial Of The Safety, Toleration and Efficacy Of Lasofoxifene 0.25 Mg/D and Raloxifene 60Mg/D For The Prevention Of Bone Loss In Postmenopausal Women
Brief Title: Comparison of Raloxifene and Lasofoxifene - A Randomized, Blinded Study of These Drugs and Placebo on Bone Loss
Acronym: CORAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Director, Project Management, Ligand Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A2181030
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Lasofoxifene; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Lasofoxifene 0.25 mg (Experimental): lasofoxifene 0.25 mg/day
  Interventions: Drug: lasofoxifene
- raloxifene (Active Comparator): raloxifene 60 mg/day
  Interventions: Drug: raloxifene
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lasofoxifene — lasofoxifene 0.25mg
  Arms: Lasofoxifene 0.25 mg
Drug: raloxifene — raloxifene 60 mg/day
  Arms: raloxifene
Drug: Placebo — 0 mg/day
  Arms: Placebo

SUMMARY:
To compare the effects of 2 years of lasofoxifene treatment with 2 years of raloxifene 60 mg/day use and 2 years of placebo use on bone mineral density (BMD) of the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with low bone density (osteopenia) and screening labs, pelvic ultrasound, mammogram without significant findings

Exclusion Criteria:

* Presence of metabolic bone disease, fractures, blood clots, or recent cancer.
* Any use of selective estrogen receptor modulators, investigational drugs, or recent use of osteoporosis treatments, certain hormones, or medication for blood clots or seizures.

Ages: 48 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2003-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Spine BMD after 2 years | 2 years
  Lumbar Spine Bome Mineral Density

SECONDARY OUTCOMES:
Hip BMD and LDL-C after 2 years, vaginal pH and Maturation Index after 1 year | Hip BMD= 24 months, LDL-C= 24 months, vaginal pH= 24 months, vaginal epithelial parabasel cells= 12 months
  Direct low density lipoprotein cholesterol (LDL-C) at 24 months, vaginal pH at 24 months, vaginal epithelial parabasal cells at 12 months, and total hip BMD at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (52):
  - Pfizer Investigational Site, Albany, California
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Brandon, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Key Largo, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Leesburg, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Gaithersberg, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Arden Hills, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Monessen, Pennsylvania
  - Pfizer Investigational Site, Mosessen, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Wyomissing, Pennsylvania
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Cordova, Tennessee
  - Pfizer Investigational Site, Germantown, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, American Fork, Utah
  - Pfizer Investigational Site, Pleasant Grove, Utah
  - Pfizer Investigational Site, Provo, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Chesapeake, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Seattle, Washington